CLINICAL TRIAL: NCT03791554
Title: Clinical Efficacy of Laterally Closed Tunnel With Subepithelial Connective Tissue Graft Versus Tunneling Technique With Subepithelial Connective Tissue Graft in Isolated Recession Type 2; Randomized Clinical Trial
Brief Title: Laterally Closed Tunnel VS Tunneling Technique in Recession Type 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yahya Hassan El Banna Amer, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Perio2414
Record Dates: First submitted 2018-12-15; First posted 2019-01-02 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Gingival Recession
Keywords: tunneling; laterally closed tunnel; gingival recession; recession type 2
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Its a randomised clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A : Lateral closed Tunnel (Active Comparator): Laterally closed tunnel procedure with subepithelial connective tissue graft (sCTG) After local anesthesia, root planing will be performed. Recession defect - a tunneling technique will be prepared using sulcular incision is made through the gingival margin and extends post the mucogingival line leaving the interdental papilla intact.
  • Recipient site; Using either single or mattress sutures, the graft will be pulled and fixed mesially and distally at the inner aspect of the pouch. The graft will be adapted to the CEJ by means of a sling suture. Margins of the pouch will be pulled together over the graft and sutured with interrupted sutures to accomplish tension-free complete or partial coverage of the graft as well as the denuded root surface.
  Interventions: Procedure: Group A (Lateral closed tunnel subepithelial CT graft)
- Group B : Tunneling (Active Comparator): Tunnel procedure with subepithelial connective tissue graft (sCTG) - Control:
  At the recipient site (recession defect): a tunneling technique will be prepared using sulcular incision is made through the gingival margin and extends post the mucogingival line leaving the interdental papilla intact.
  Then the graft is placed and secured in the recipient site. The flap is displaced to be in a coronal position using a sling suture with no suturing to approximate the margins together.
  Interventions: Procedure: Group B (Tunnel procedure with subepithelial CT graft)

INTERVENTIONS:
Procedure: Group A (Lateral closed tunnel subepithelial CT graft) — Subepithelial connective tissue graft (autogenous graft) will be harvested from the palate by Single incision technique to be used with the adjacent teeth to treating gingival recession with edges of the recession sutured together after placing connective tissue graft
  Arms: Group A : Lateral closed Tunnel
Procedure: Group B (Tunnel procedure with subepithelial CT graft) — Subepithelial connective tissue graft (autogenous graft) will be harvested from the palate by Single incision technique to be used with the prepared tunnel to treating gingival recession
  Other Names: Autogenous sCTG will be used with tunnel procedure
  Arms: Group B : Tunneling

SUMMARY:
This study aims to assess the effect of tunneling technique with subepithelial connective tissue graft versus tunneling technique with laterally closed tunnel in treatment of recession type 2 defect.Few randomized clinical trial has been involved with recession type 2 defects treated with tunneling technique and coronal advanced flap.

DETAILED DESCRIPTION:
Tunneling with subepithelial connective tissue graft:

At the recipient site (recession defect):

After scaling and root planning. A sulcular incision is made through the gingival margin and extends post the mucogingival line leaving the interdental papilla intact.

At donor site (palate):

A connective tissue graft is harvested from the palate after administration of local anesthesia using a partial thickness flap which will be raised with single incision.

Then the graft is placed and secured in the recipient site using suture. The flap is displaced to be in a coronal position using a suture.

Tunneling technique with the laterally closed tunnel):

After local anesthesia, root planing of the exposed root surface will be performed. An intrasulcular incisions will be made creating a tunnel extending to the mucogingival line and mesial and distal recession defects while keeping the interdental papilla intact as well as not perforating the flap.

* Donor SCTG Subsequently, a palatal SCTG will be harvested by means of the single incision technique with immediate closure of the donor site.
* Recipient site; Using either single or mattress sutures, the SCTG will be pulled and fixed mesially and distally at the inner aspect of the pouch. The graft will be adapted to the CEJ by means of a sling suture. Finally, the margins of the pouch will be pulled together over the graft and sutured with interrupted sutures to accomplish tension-free complete or partial coverage of the graft as well as the denuded root surface.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.
* Patients with healthy systemic condition
* Buccal recession defects with recession type 2 defects.
* Clinical indication and/or patient request for recession coverage.
* O'Leary index less than 20%

Exclusion Criteria:

* Pregnant females.
* Smokers as it is a contraindication for any plastic periodontal surgery
* Unmotivated, uncooperative patients with poor oral hygiene
* Patients with habits that may compromise the longevity and affect the result of the study as alcoholism or para-functional habits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Reduction Recession Depth | 6 month
  recession depth measured from CEJ to the gingival margin in a cross-section at the central buccal site.

SECONDARY OUTCOMES:
Gingival recession depth. | 6 month
  Measured as the distance between the gingival margin and the mucogingival junction
Gingival recession width | 6 month
  Measured as the distance between the gingival margin adjacent to the defect
Root coverage esthetic score (RES) | 6 month
  system used to evaluated five variables 6 months gingival margin (GM), marginal tissue contour (MTC), soft tissue texture (STT), MGJ alignment, and gingival color (GC).
Probing depth | 6 month
  Measured from the gingival margin to the bottom of the gingival sulcus
Clinical attachment level | 6 month
  Measured from the CEJ to the bottom of the gingival sulcus.
Width of keratinized tissue | 6 month
  Measured as the distance between the gingival margin and the mucogingival junction
Gingival thickness | 6 month
  The measurement of Gingival tissue thickness is performed 2 mm apical from the gingival margin.
Post-operative pain | 2 weeks
  Visual Analogue Scale (VAS) with numbers from 0 to 10 ('no pain' to 'worst' pain imaginable)
Post-Surgical Patient Satisfaction Questionnaire | 6 month
  A 3-item questionnaire is asked and the patients shall use a 7-point answer scale. The answers were given on a 7-point scale ranging from 1 ''not at all'' to 7 ''very likely''
Percentage complete root coverage | 6 month
  (Preoperative vertical recession -- Postoperative vertical recession/preoperative vertical recession) x 100

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, PhD, Study Chair — Cairo University; Hani El-Nahass, PhD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Almanyal , Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
I will check with my Study Chair

REFERENCES:
- [Background] Agudio G, Nieri M, Rotundo R, Cortellini P, Pini Prato G. Free gingival grafts to increase keratinized tissue: a retrospective long-term evaluation (10 to 25 years) of outcomes. J Periodontol. 2008 Apr;79(4):587-94. doi: 10.1902/jop.2008.070414. PMID 18380550
- [Background] Aroca S, Keglevich T, Nikolidakis D, Gera I, Nagy K, Azzi R, Etienne D. Treatment of class III multiple gingival recessions: a randomized-clinical trial. J Clin Periodontol. 2010 Jan;37(1):88-97. doi: 10.1111/j.1600-051X.2009.01492.x. Epub 2009 Nov 30. PMID 19968743
- [Background] Baldi C, Pini-Prato G, Pagliaro U, Nieri M, Saletta D, Muzzi L, Cortellini P. Coronally advanced flap procedure for root coverage. Is flap thickness a relevant predictor to achieve root coverage? A 19-case series. J Periodontol. 1999 Sep;70(9):1077-84. doi: 10.1902/jop.1999.70.9.1077. PMID 10505811
- [Background] Cairo F, Nieri M, Cincinelli S, Mervelt J, Pagliaro U. The interproximal clinical attachment level to classify gingival recessions and predict root coverage outcomes: an explorative and reliability study. J Clin Periodontol. 2011 Jul;38(7):661-6. doi: 10.1111/j.1600-051X.2011.01732.x. Epub 2011 Apr 20. PMID 21507033
- [Background] Cairo F, Rotundo R, Miller PD, Pini Prato GP. Root coverage esthetic score: a system to evaluate the esthetic outcome of the treatment of gingival recession through evaluation of clinical cases. J Periodontol. 2009 Apr;80(4):705-10. doi: 10.1902/jop.2009.080565. PMID 19335093
- [Background] Cortellini P, Tonetti M, Baldi C, Francetti L, Rasperini G, Rotundo R, Nieri M, Franceschi D, Labriola A, Prato GP. Does placement of a connective tissue graft improve the outcomes of coronally advanced flap for coverage of single gingival recessions in upper anterior teeth? A multi-centre, randomized, double-blind, clinical trial. J Clin Periodontol. 2009 Jan;36(1):68-79. doi: 10.1111/j.1600-051X.2008.01346.x. Epub 2008 Nov 20. PMID 19046326
- [Background] Dominiak M, Gedrange T. New perspectives in the diagnostic of gingival recession. Adv Clin Exp Med. 2014 Nov-Dec;23(6):857-63. doi: 10.17219/acem/27907. PMID 25618109
- [Background] Edel A. Clinical evaluation of free connective tissue grafts used to increase the width of keratinised gingiva. 1974. Periodontal Clin Investig. 1998 Spring;20(1):12-20. No abstract available. PMID 9663118
- [Background] Esteibar JR, Zorzano LA, Cundin EE, Blanco JD, Medina JR. Complete root coverage of Miller Class III recessions. Int J Periodontics Restorative Dent. 2011 Jul-Aug;31(4):e1-7. PMID 21837295
- [Background] Kassab MM, Cohen RE. The etiology and prevalence of gingival recession. J Am Dent Assoc. 2003 Feb;134(2):220-5. doi: 10.14219/jada.archive.2003.0137. PMID 12636127
- [Background] Khuller N. Coverage of gingival recession using tunnel connective tissue graft technique. J Indian Soc Periodontol. 2009 May;13(2):101-5. doi: 10.4103/0972-124X.55838. PMID 20407659
- [Background] Langer B, Langer L. Subepithelial connective tissue graft technique for root coverage. J Periodontol. 1985 Dec;56(12):715-20. doi: 10.1902/jop.1985.56.12.715. PMID 3866056
- [Background] Miller PD Jr. A classification of marginal tissue recession. Int J Periodontics Restorative Dent. 1985;5(2):8-13. No abstract available. PMID 3858267
- [Background] Nordland WP, Tarnow DP. A classification system for loss of papillary height. J Periodontol. 1998 Oct;69(10):1124-6. doi: 10.1902/jop.1998.69.10.1124. PMID 9802711
- [Background] Raetzke PB. Covering localized areas of root exposure employing the "envelope" technique. J Periodontol. 1985 Jul;56(7):397-402. doi: 10.1902/jop.1985.56.7.397. PMID 3894614
- [Background] Sculean A, Allen EP. The Laterally Closed Tunnel for the Treatment of Deep Isolated Mandibular Recessions: Surgical Technique and a Report of 24 Cases. Int J Periodontics Restorative Dent. 2018 Jul/Aug;38(4):479-487. doi: 10.11607/prd.3680. PMID 29889911
- [Background] Shah R, Thomas R, Mehta DS. Recent modifications of free gingival graft: A case series. Contemp Clin Dent. 2015 Jul-Sep;6(3):425-7. doi: 10.4103/0976-237X.161910. PMID 26321849
- [Background] Smith RG. Gingival recession. Reappraisal of an enigmatic condition and a new index for monitoring. J Clin Periodontol. 1997 Mar;24(3):201-5. doi: 10.1111/j.1600-051x.1997.tb00492.x. PMID 9083906
- [Background] Sullivan HC, Atkins JH. Free autogenous gingival grafts. I. Principles of successful grafting. Periodontics. 1968 Jun;6(3):121-9. No abstract available. PMID 5240496
- [Background] Zabalegui I, Sicilia A, Cambra J, Gil J, Sanz M. Treatment of multiple adjacent gingival recessions with the tunnel subepithelial connective tissue graft: a clinical report. Int J Periodontics Restorative Dent. 1999 Apr;19(2):199-206. PMID 10635186
- [Background] Zucchelli G, Mounssif I. Periodontal plastic surgery. Periodontol 2000. 2015 Jun;68(1):333-68. doi: 10.1111/prd.12059. PMID 25867992